CLINICAL TRIAL: NCT01116349
Title: Diaphyseal Fractures of the Humerus: A Prospective Cohort Study Comparing the Conservative Treatment and the Surgical Treatment.
Brief Title: Conservative Treatment Versus the Surgical Treatment of Diaphyseal Fractures of Humerus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties to recruit participants A similar Canadian multicentric study started at about the same.
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Principal Investigator, Pelet Stephane, Dr Stephane Pelet MD, PhD Orthopedic surgeon, Hopital de l'Enfant-Jesus
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEJ-530
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Humeral Diaphysis Fracture
Keywords: humeral diaphysis fracture; plate and screws for humeral diaphysis fracture; nailing for humerus diaphysis fracture; Hanging Support System
MeSH Terms: interventions — Bone Plates; Fracture Fixation, Intramedullary; Braces

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical treatment (Active Comparator): Patients included in the surgical group will have surgery to treat the fracture.
  Interventions: Procedure: Plate and screws or nailing
- Conservative treatment group (Active Comparator): Patients included in the conservative group will be taken to a plaster room where a Hanging Support System(HSS) brace will be installed by a qualified technician.
  Interventions: Device: Hanging Support System (HSS) brace

INTERVENTIONS:
Procedure: Plate and screws or nailing — Patients included in the surgical group will be divided into two subgroups according to the method of fixation chosen: plate and screws or nailing. Surgeries take place under general anesthesia and a prophylaxis antibiotic is administrated. The installation and the approach will be chosen by the surgeon according to his preferences. A thoraco brachial brace is placed on the patient at the end of the intervention and it remains in place for a period of 5 to 10 days (patient comfort). A gradual mobilization of the elbow and shoulder will be initiated by the patient at home. The addition of physical therapy will be decided by the surgeon and noted down accordingly.
  Arms: Surgical treatment
Device: Hanging Support System (HSS) brace — Patients included in the conservative group will be taken to a plaster room where the HSS brace will be installed by a qualified technician. Advice will be provided for the care, personal hygiene and clothing. The brace will be kept for a period of 6 to 12 weeks depending on the degree of healing of fracture. The maintenance of the proximal part (Brace) may be recommended by the surgeon. The mobilization will begin with exercises at home and whether the patient does physical therapy or not is the surgeon's choice.
  Arms: Conservative treatment group

SUMMARY:
The fracture of the humeral diaphysis is a condition that represents 2% of all fractures. The conservative treatment of diaphyseal fractures of the humerus has long been considered the only option and the surgical treatment was primarily reserved for displaced fractures with no contact of bone ends. However, for a few years there has been an upsurge of indications for the surgical treatment of diaphyseal fractures.

The purpose of this study is to compare the functional outcomes and the quality of life of surgically treated patients versus those who undergo a conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years
* Fracture of the humeral diaphysis
* Recent fracture (14 days or less)
* Closed fracture
* Signing of consent form

Exclusion Criteria:

* Segmental fracture of the humerus
* Fracture with proximal or distal intra articular extension
* Open fracture
* Polytrauma
* Floating elbow or shoulder
* Pathological fracture
* Simultaneous fracture of both humerus
* Associated vascular disease
* Severe neuromuscular disorders such as Parkinson, hemiparesis, myasthenia gravis, muscular dystrophy, etc. ...
* medical contraindication to surgery
* severe central neurological disease disabling patient to fill in questionnaires (senile dementia, Alzheimer's, etc ...
* Male or female unable to consent
* Any other condition which prevents the assessor from fully monitoring the patient during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Function and quality of life on DASH scale | 6 months after treatment
  The function and quality of life are measured using the DASH scale six months after treatment.

SECONDARY OUTCOMES:
DASH score | 6 months after treatment
  The function and quality of life are measured using the DASH scale 6 months after treatment.
Return to professional activities | 3 months after treatment
  It will be determined in days after surgery, to rates of 50% and 100% of the usual workload.
SF-36 score | 6 months after treatment
  This score will help validate the impact on quality of life of both types of treatment. It includes 36 items asking about the recent quality of life. This will also enable better understanding of the impact in real time on the functional level.
DASH score | 12 months after treatment
  The function and quality of life are measured using the DASH scale 12 months after treatment.
SF-36 score | 12 months after treatment
  This score will help validate the impact on quality of life of both types of treatment. It includes 36 items asking about the recent quality of life. This will also enable better understanding of the impact in real time on the functional level.
Proportion of additional surgeries | 12 months after surgery
  The evaluation of the rate of complications such as infection, implant removal, non-union, implant failure or malunion which necessitate additional surgery.
Radiological loss of reduction | 2 weeks after treatment
  The main observed displacements occur in varus and are measured on an AP view of the humerus. Initial displacements are tolerated up to 20 degrees in varus and in flexion.
  We measure the proportion of patients who experienced worsening of the deformity of more than 5 degrees on both levels.
Radiological loss of reduction | 6 weeks after treatment
  The main observed displacements occur in varus and are measured on an AP view of the humerus. Initial displacements are tolerated up to 20 degrees in varus and in flexion.
  We measure the proportion of patients who experienced worsening of the deformity of more than 5 degrees on both levels.
Radiological loss of reduction | 12 weeks after treatment
  The main observed displacements occur in varus and are measured on an AP view of the humerus. Initial displacements are tolerated up to 20 degrees in varus and in flexion.
  We measure the proportion of patients who experienced worsening of the deformity of more than 5 degrees on both levels.
Radiological loss of reduction | 6 months after treatment
  The main observed displacements occur in varus and are measured on an AP view of the humerus. Initial displacements are tolerated up to 20 degrees in varus and in flexion.
  We measure the proportion of patients who experienced worsening of the deformity of more than 5 degrees on both levels.
Union rate | 12 weeks after treatment
  The union is defined by the presence of a strong radiological callus associated with lack of pain at the fracture site. The humerus unifies in an average of three months. It is considered non-union if it is not unified after six months, and it is classified as delayed union between 3 and 6 months.
  The rates will be presented by the number of patients with non-union in each group.
Union rate | 6 months after treatment
  The union is defined by the presence of a strong radiological callus associated with lack of pain at the fracture site. The humerus unifies in an average of three months. It is considered non-union if it is not unified after six months, and it is classified as delayed union between 3 and 6 months.
  The rates will be presented by the number of patients with non-union in each group.
Rates of complication | within the first year following treatment
  The main complications recognized in the treatment of humerus fractures are: infection, nerve damage, malunion and non-unions. Each complication will be recorded and reported.
Pain on visual analogue pain scale (VAS) | 2 weeks after treatment
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full of numbers 1 to 10.
Pain on VAS | 6 weeks after treatment
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full of numbers 1 to 10.
Pain on VAS | 12 weeks after treatment
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full of numbers 1 to 10.
Pain on VAS | 6 months after treatment
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full of numbers 1 to 10.
Pain on VAS | 12 months after treatment
  The measure will be carried out using a suitable rule designed for this type of measurement, counting only full of numbers 1 to 10.
Measurement of range of motion of the shoulder | 2 weeks after treatment
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180°), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60°).
Measurement of range of motion of the shoulder | 6 weeks after treatment
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180°), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60°).
Measurement of range of motion of the shoulder | 12 weeks after treatment
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180°), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60°).
Measurement of range of motion of the shoulder | 6 months after treatment
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180°), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60°).
Measurement of range of motion of the shoulder | 12 months after treatment
  Using a goniometer, we will measure the bending (normal value 180 °), abduction (180°), external rotation in the scapular plane (90 °) and internal rotation in the plane scapula (60°).
Measurement of range of motion of the elbow | 2 weeks after treatment
  Using a goniometer, we will measure the bending (normal value 140 °), extension (normal value 0 °), pronation (normal value 80 °) and supination (normal value 80 °).
Measurement of range of motion of the elbow | 6 weeks after treatment
  Using a goniometer, we will measure the bending (normal value 140 °), extension (normal value 0 °), pronation (normal value 80 °) and supination (normal value 80 °).
Measurement of range of motion of the elbow | 12 weeks after treatment
  Using a goniometer, we will measure the bending (normal value 140 °), extension (normal value 0 °), pronation (normal value 80 °) and supination (normal value 80 °).
Measurement of range of motion of the elbow | 6 months after treatment
  Using a goniometer, we will measure the bending (normal value 140 °), extension (normal value 0 °), pronation (normal value 80 °) and supination (normal value 80 °).
Measurement of range of motion of the elbow | 12 months after treatment
  Using a goniometer, we will measure the bending (normal value 140 °), extension (normal value 0 °), pronation (normal value 80 °) and supination (normal value 80 °).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Pelet, MD, PhD, Principal Investigator — Hôpital de l'Enfant-Jésus
Locations (2):
- Canada (2):
  - CHA-Pavillon Enfant-Jésus, Québec, Quebec
  - Hôpital l'Enfant-Jésus, Québec, Quebec